CLINICAL TRIAL: NCT00638521
Title: Trauma and Sepsis Induced Changes in Immune-cell Membrane Receptor Trafficking
Brief Title: Immune-cell Membrane Trafficking
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Joseph Cuschieri, Study Principal Investigator, University of Washington
Other Study IDs: 31888-A; GM078054-01 (Other: National Institute of General Medical Sciences (NIGMS))
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Severe Trauma
Keywords: lipids; proteins; membrane; lipid raft
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Organ failure following trauma is a leading cause of morbidity and mortality. It appears that the development of organ failure is a direct result of an altered immune response. This altered response results in the production of circulating factors in the blood that causes direct injury to the injured patients' organs. The mechanism in which this altered immune response occurs is unknown. Based on work we have performed in our laboratory, we believe that this response is initiated on the cell membrane of particular immune cells known as macrophages. Although the cell membrane may appear uniform, it is not. The membrane is composed of specific segments that allow proteins to associate with each other forming receptors that are required for immune cell activation. These specific membrane components are composed of various lipids and cholesterol, and have been termed lipid rafts. Based on our laboratory work it appears that these lipid rafts can be altered following injury. In particular both the lipid and protein content within these raft segments may be altered allowing immune cells to become active leading to the production of factors that directly injure normal cells and organs. Thus, we plan to examine if these laboratory findings can be seen in patients suffering from trauma who develop clinical organ failure at Harborview Medical Center. If this is accomplished, this data will lead to the development of both prognostic and therapeutic interventions for the optimal care of injured patient

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older, blunt or penetrating trauma and
* one or more of the following: systolic blood pressure less than 90 mmHg at the scene or within one hour of arrival to the Emergency Department, 2) base deficit ≥ -6 within one hour of admission, 3) ISS greater than 25, or 4) more than 6 units of blood transfused in the first 12 hours.-

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessment of protein and lipid changes in immune cells following severe injury | 5/08 to 8/12

SECONDARY OUTCOMES:
Assessment of severe injury effect on plasma and cellular lipid content | 5/08 to 8/12

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cuschieri, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States